CLINICAL TRIAL: NCT02915458
Title: Predictive Analysis Software for Successful Weaning From Ventilator of Patients in Critical Condition
Brief Title: Predictive Analysis Software for Successful Weaning From Ventilator of Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Lun Lo, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 104-6531B
Record Dates: First submitted 2016-07-19; First posted 2016-09-27 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Weaning Failure
Keywords: Weaning; Mechanical ventilation; synchrosqueezing transform

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Making a weaning decision for a patient on a mechanical ventilator is an important clinical issue. The most common index to predict successful weaning is the rapid shallow breathing index (RSBI), however, the accuracy of RSBI to predict successful weaning have been questioned.

The investigators proposed a new mathematical model and algorithm, called WIN, which capture the essential feature of the variability ruling the physiological dynamics to provides better perdition to wean than RSBI.

DETAILED DESCRIPTION:
Making a weaning decision for a patient on a mechanical ventilator is an important clinical issue.

It is thus important to decide accurately when patients can be weaned from the ventilator. To increase the weaning success, the present common practice is to conduct spontaneous breathing trials to get physiological signals that may provide the information about capacity of successful weaning. The most common index is the rapid shallow breathing index (RSBI), however, the accuracy of RSBI to predict successful weaning have been questioned. Weaning failure usually results from a complex interplay of multiple factors. Thus, predictors targeting a single pathophysiologic mechanism tend to be unreliable for heterogeneous abnormalities.

The investigators proposed a new mathematical model and algorithm, which capture the essential feature of the variability ruling the physiological dynamics. Through the modern adaptive signal processing techniques, the investigators develop an index called WIN, which is evaluated from the 5 minutes continuous physiological signal and provides better perdition to wean than RSBI in a retrospective analysis. In this study, the investigators evaluate the predictive power of WIN and RSBI prospectively in patients undergoing weaning prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mechanical ventilation via an endotracheal tube (oral endotracheal tube or tracheostomy tube) for >24 hours; 2. Patients are concomitant with presence of the following criteria of ready be weaned, a spontaneous breathing trial (SBT) will then be evaluated by 120-min T-piece:

1. clear improvement of the condition that led to mechanical ventilation;
2. no acute pulmonary or neuromuscular disease or signs of increased intracranial pressure;
3. conscious and lying on a bed with the upper body elevated to a 30◦ angle
4. adequate oxygenation (PaO2 ≥ 60mmHg and fraction of inspired oxygen inspired oxygen fraction (FiO2) ≤ 40% with positive end expiratory pressure (PEEP) ≤ 8cm H2O, or PaO2 /FiO2 >150 mmHg);
5. no significant respiratory acidosis, PaCO2<50mmHg, or increasing <10% for patients with chronic CO2 retention.
6. stable cardiovascular status (Heat beat ≤140/min, systolic blood pressure 90-160mmHg);
7. no requirement for vasopressive or inotropic dugs≥ 8 hours;
8. no intravenous sedatives during the previous 24 hours;
9. ability to cough while suction;
10. afebrile with ≤ 38◦ C temperature.
11. negative cuff leakage test: >110ml or >12%

Exclusion Criteria:

1. Presence of tracheostomy
2. Home ventilation prior to ICU admission
3. Decision not to re-intubate or withdrawal of care anticipated
4. Further surgery requiring sedation planned next 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with mechanical ventilation via an endotracheal tube (oral endotracheal tube or tracheostomy tube) for >24 hours;
  2. Patients are ready be weaned to performed a spontaneous breathing trial by 120-min T-piece.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Successful weaning from mechanical ventilation | up to 72 hours
  The patients could breath by themselves after extubation without any ventilator assistance for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Lun Lo, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu HT, Talmon R, Lo YL. Assess sleep stage by modern signal processing techniques. IEEE Trans Biomed Eng. 2015 Apr;62(4):1159-1168. doi: 10.1109/TBME.2014.2375292. Epub 2014 Nov 26. PMID 25438301
- [Background] Wu HT, Hseu SS, Bien MY, Kou YR, Daubechies I. Evaluating physiological dynamics via synchrosqueezing: prediction of ventilator weaning. IEEE Trans Biomed Eng. 2014 Mar;61(3):736-44. doi: 10.1109/TBME.2013.2288497. Epub 2013 Nov 4. PMID 24235294